CLINICAL TRIAL: NCT05635318
Title: Quantitative EEG Neurofeedback as an Add-on Therapy For Attention-deficit Hyperactivity Disorder (ADHD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Emad Eldeen Mahmoud, Mohamed Emad Eldaly, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QEEG-NF for ADHD
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Dosage Forms; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Placebo Comparator): Group A including ADHD patients who will be treated according to The American academy of Pediatrics Guidelines with FDA-approved medications
  Interventions: Drug: FDA approved medications for ADHD
- Group B (Active Comparator): Group A including ADHD patients who will be treated according to The American academy of Pediatrics Guidelines with FDA-approved medications plus Quantitative EEG Neurofeedback
  Interventions: Device: FDA approved medications for ADHD plus Quantitative EEG Neurofeedback

INTERVENTIONS:
Device: FDA approved medications for ADHD plus Quantitative EEG Neurofeedback — A mathematical approach to analyzing EEG data, called quantitative electroencephalography (qEEG), can be used to develop a visual map of the type and location of brain waves or rhythms. Other more specific wave patterns, such as event-related potentials, can also be seen in the EEG.NF converts signals such as EEG into visual or auditory information, and then subjects selectively enhance or inhibit certain components through training. There are three common NF protocols for ADHD: theta/beta training, sensorimotor rhythm (SMR) training, and slow cortical potentials (SCP) training.
  Other Names: Drugs + QEEG-NF
  Arms: Group B
Drug: FDA approved medications for ADHD — Ritalin (methylphenidate HCl); Ritalin LA, Ritalin SR Strattera (atomoxetine HCl)
  Other Names: Drugs
  Arms: Group A

SUMMARY:
Attention deficit/hyperactivity disorder (ADHD) is a common neurological disorder in children, mainly manifesting as attention deficit, excessive hyperactivity, and impulsivity. It is a chronic condition that affects millions of children and often continues into adulthood.

The prevalence of ADHD in the worldwide is approximately 5%, predominantly occurring in boys, and more than half of patients continue to experience symptoms into adulthood. Children with ADHD have moral disorders and learning difficulties, and these factors will seriously affect their academic achievements and familial and social relationships; thus, treatment is necessary.

Currently, the treatment for ADHD is usually pharmacological intervention, such as methylphenidate, Atomoxetine…. etc. However, research has suggested that pharmacological intervention has side effects on nervous system development in children, and the long-term efficacy is uncertain. In recent years, the efficacy of neurofeedback (NF) therapy, as a type of biofeedback method, has been proven in many diseases, such as mild cognitive impairment, epilepsy, and autism, depression, and anxiety.

NF converts signals such as EEG into visual or auditory information, and then subjects selectively enhance or inhibit certain components through training. There are three common NF protocols for ADHD: theta/beta training, sensorimotor rhythm (SMR) training, and slow cortical potentials (SCP) training. This study adopts the theta/beta NF protocol. As a promising nonpharmacological alternative treatment for ADHD, the efficacy of NF has been proven in many studies.

The use of quantitative EEG neurofeedback as an add-on therapy can be markedly beneficial to shorten the period of pharmacological treatment and with minimal side effects.

DETAILED DESCRIPTION:
Attention deficit/hyperactivity disorder (ADHD) is a common neurological disorder in children, mainly manifesting as attention deficit, excessive hyperactivity, and impulsivity. It is a chronic condition that affects millions of children and often continues into adulthood. ADHD includes a combination of persistent problems, such as difficulty sustaining attention, hyperactivity, and impulsive behavior. Based on the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV), the American Psychiatric Association has divided ADHD into three subtypes: predominantly inattention (ADHD-I), predominantly hyperactive-impulsive (ADHD-HI) and a combination of both (ADHD-C) (1) The prevalence rate of ADHD in the worldwide is approximately 5%, predominantly occurring in boys, and more than half of patients continue to experience symptoms into adulthood (2). Most children with ADHD have moral disorders and learning difficulties, and these factors will seriously affect their academic achievements and familial and social relationships; thus, prompt treatment is necessary. (3) Historically, conventional EEG has added little to the understanding of childhood psychiatric disorders, other than to rule out epilepsy or space occupying lesions. However, the advent of computerized, quantitative methods, together with new neuroimaging techniques as brain sources localization and the availability of normative databases both of normal subjects and of subjects with definite pathologies has greatly enhanced the clinical application in neurodevelopmental disorders. Furthermore, in these past years, it has become more and more apparent that groups of patients with neuropsychiatric disorders, who meet symptom based diagnostic criteria for specific disorders (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition [DSM-IV] or International Classification of Diseases, 10th Revision [ICD-10]) have varied responses to treatment, despite their relatively homogeneous clinical presentation. Using clinical diagnosis, the "treatment of choice" leads to a positive response approximately 60% of the time. (4) This poor response rate suggests heterogeneity within these relatively homogeneous clinical populations. In this direction, the term personalized medicine is becoming more and more common, a medical procedure that separates patients into different groups based on their electrophysiological profiles and predicted response to the quantitative EEG. This has allowed the study of single subjects and to customize health care, with decisions and treatments tailored to each individual patient, as well as improvement of knowledge of the pathophysiological mechanisms of specific diseases.

Currently, the treatment for ADHD is usually pharmacological intervention, such as methylphenidate, Atomoxetine…. etc. However, research has suggested that pharmacological intervention has side effects on nervous system development in children, and the long-term efficacy is uncertain. In recent years, the efficacy of neurofeedback (NF) therapy, as a type of biofeedback method, has been proven in many diseases, such as mild cognitive impairment, epilepsy, and autism, depression and anxiety. Stemming from Skinner's operant conditioned reflexes theory, NF is to enable individuals to actively control and adjust according to their own EEG changes to achieve a certain criterion and finally achieve the purpose of regulating brain function. (5) Neurofeedback (also called neurotherapy or electroencephalogram [EEG] biofeedback) is a type of biofeedback that uses conditioning to train people to improve regulation of their brain-wave patterns by providing them with real-time video/audio information about their brain's electrical activity measured from scalp electrodes. In effect, the conditioning is based on feedback given to the patient that is contingent on the patient's EEG pattern.

First described qualitatively as "brain waves" on the EEG by Hans Berger in 1924, the electrical activity of the brain was thought to reflect changes in the brain's functional state while awake or asleep, or to denote brain diseases such as epilepsy. (6) EEG activity, characterized in terms of rhythmic activity measured in hertz (Hz, the number of waves per second), is divided into specifically named frequency bands, corresponding to functional activity and arousal state: the delta band corresponds to slow-wave sleep state (up to 4 Hz), Theta to a drowsy/inattentive state (4-8 Hz), alpha to a relaxed/wakeful/alert state (8-12 Hz), and beta to an active/attentive state (12-30 Hz).Most of the brain electrical activity occurs in the 1- to 20-Hz range.

Within each band, there are recognizable functionally significant rhythms. For example, a specific type of low beta activity (12-15 Hz) observed in the sensorimotor cortex is called the sensorimotor rhythm. The amplitude of the sensorimotor rhythm is higher when the sensory-motor areas are inactive (eg, during immobile states) and decreases when those areas are activated (eg, during motor tasks). Therefore, the amplitude of the sensorimotor rhythm is a measure of sensory-motor inhibition; that is, higher amplitude when the "brake is on" and lower when the "brake is off." A mathematical approach to analyzing EEG data, called quantitative electroencephalography (qEEG), can be used to develop a visual map of the type and location of brain waves or rhythms. Other more specific wave patterns, such as event-related potentials, can also be seen in the EEG. Event-related potentials are electrical representations associated with sensory and cognitive processing occurring in response to a stimulus or event. (7) Slow cortical potentials (SCPs) are one specific group of event-related potentials. They are slow event-related direct-current shifts of the EEG that correspond to the excitation threshold of large cortical cell assemblies. (8,9) Shifts in the positive direction indicate an increase of the excitation threshold and a corresponding inhibition of activation, whereas shifts in the negative direction, called the contingent negative variation, reflect a reduction of the excitation threshold, and represent cognitive preparation and increased cortical activation of a network. (8,10) The classical conditioning of human EEG was first shown in the mid- 1930s, when researchers trained human subjects to block a wave. (7,8) Operant conditioning, in which EEG-derived information is used as instant feedback to the patient in realtime, was first used to alter the human EEG in the 1960s (11,12,13) Since the 1960s, mainly using operant conditioning, there has been a significant increase in the clinical application of NF to several neuropsychiatric conditions, including ADHD, LD, developmental disabilities, cognitive/memory enhancement, epilepsy, traumatic brain injury, stroke, alcoholism, substance abuse, antisocial personality, autism, anxiety, depression, insomnia, and migraines.(14) There has also been a significant increase, especially in the 21st century, in the number of published research and dissertation studies TYPES OF NEUROFEEDBACK

There are 7 types of NF, Hammond (15) defines their use for various disorders:

1. The traditional and most frequently used is Frequency/Power NF, and it is the NF method usually meant by the general term "neurofeedback." This technique typically entails the use of 2 to 4 surface electrodes and is sometimes called "surface neurofeedback." Developed in the 1960s to change the amplitude or speed of specific brain waves in particular brain locations, it is used to treat ADHD, anxiety, insomnia, and LD.
2. Slow Cortical Potential Neurofeedback (SCP-NF) modifies the direction (positive or negative) of slow cortical potentials and has been used to treat epilepsy, migraines, and ADHD.
3. Low-Energy Neurofeedback System (LENS), developed in 1992, is a passive type of NF involving delivery of a very weak electromagnetic signal to change a patient's brain waves while the patient is motionless and has their eyes closed; it has been used to treat traumatic brain injury, fibromyalgia, anger, restless legs syndrome, ADHD, anxiety, depression, and insomnia.
4. Hemoencephalographic (HEG) Neurofeedback, developed in 1994, provides feedback about cerebral blood flow to treat migraine.
5. Live Z-score Neurofeedback, developed in 1998, involves the continuous comparison of multiple variables of brain electrical activity (eg, power, asymmetries, phase-lag, coherence) to a normative database to give moment-to-moment feedback; it has been used to treat insomnia.
6. Low-Resolution Electromagnetic Tomography (LORETA) was developed in 1994 to treat depression, addictions, and obsessive-compulsive disorder. LORETA involves the use of 19 electrodes that are used to monitor phase, power, and coherence
7. The most recent type of NF, developed in 2003, is functional magnetic resonance imaging (fMRI) NF, which allows patients to regulate their brain activity based on feedback of activity from deep subcortical areas of the brain.

NF has been suggested for the treatment of ADHD because research indicates that many patients with ADHD have more slow-wave (especially Theta, 3.5-8 Hz) power and less beta (12-20 Hz) power, especially in the central and frontal regions, as well as reduced cortical negativity (ie, a deviance in contingent negative variation) during cognitive preparation. These brain-wave patterns probably reflect under arousal of the central nervous system associated with the core ADHD symptoms of inattention, hyperactivity, and impulsivity. The goal of this treatment is to reverse these functional characteristics of abnormal CNS physiology by countering the physiological under arousal associated with ADHD.

NF converts signals such as EEG into visual or auditory information, and then subjects selectively enhance or inhibit certain components through training. There are three common NF protocols for ADHD: theta/beta training, sensorimotor rhythm (SMR) training, and slow cortical potentials (SCP) training. (16) This study adopts the theta/beta NF protocol. As a promising nonpharmacological alternative treatment for ADHD, the efficacy of NF has been proven in many studies. Meisel et al. conducted a six-month follow-up trial that compared NF and medication in children with ADHD and discovered significant academic performance improvements in only the NF group (17). One study reported that NF can not only be used as a therapy for many neuropsychiatric disorders but also improve the emotion and cognition of healthy people (18) So the use of quantitative EEG neurofeedback as an add-on therapy can be markedly beneficial to shorten the period of pharmacological treatment and with minimal side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ADHD according to DSM-5 Criteria for ADHD Age group: 4 years up to less than 16 years

Exclusion Criteria:

* *Any patient with other neurological or psychological diseases e.g. Epilepsy, Autism, Cerebral palsy

  * Any patient in a different age group

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of ADHD manifestations | 6 months
  Greater improvement in ADHD score between group B and Group A

SECONDARY OUTCOMES:
Improvement of intelligence | 1 year
  with the diminished manifestations of ADHD, the IQ is expected to be increased

REFERENCES:
- [Background] Arns M, Drinkenburg W, Leon Kenemans J. The effects of QEEG-informed neurofeedback in ADHD: an open-label pilot study. Appl Psychophysiol Biofeedback. 2012 Sep;37(3):171-80. doi: 10.1007/s10484-012-9191-4. PMID 22446998
- [Background] Krepel N, Egtberts T, Sack AT, Heinrich H, Ryan M, Arns M. A multicenter effectiveness trial of QEEG-informed neurofeedback in ADHD: Replication and treatment prediction. Neuroimage Clin. 2020;28:102399. doi: 10.1016/j.nicl.2020.102399. Epub 2020 Aug 25. PMID 32891892